CLINICAL TRIAL: NCT00270010
Title: A Double-Blind, Placebo-Controlled Study With Open-Label Follow-up to Determine the Safety and Efficacy of Subcutaneous Doses of r-HuEPO in AIDS Patients With Anemia Induced by Their Disease and AZT Therapy
Brief Title: A Study to Evaluate the Safety and Effectiveness of Epoetin Alfa in AIDS (Acquired Immunodeficiency Syndrome) Patients With Anemia Caused Both by Their Disease and by AZT (Zidovudine, an Antiviral Drug) Given as Treatment for Their Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR005842
Record Dates: First submitted 2005-12-22; First posted 2005-12-26 (Estimated); Last update posted 2011-05-18 (Estimated); Status verified 2010-04

CONDITIONS: Anemia; Acquired Immunodeficiency Syndrome
Keywords: Anemia; AIDS; HIV; Zidovudine; Quality of Life; erythropoietin; epoetin alfa
MeSH Terms: conditions — Anemia; Acquired Immunodeficiency Syndrome | interventions — Epoetin Alfa

INTERVENTIONS:
Drug: epoetin alfa

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of epoetin alfa versus placebo for the treatment of anemia in AIDS (Acquired Immunodeficiency Syndrome) patients with anemia that is a result of this disease and zidovudine (AZT) treatment. Epoetin alfa is a genetically engineered protein that stimulates red blood cell production.

DETAILED DESCRIPTION:
It is estimated that approximately 75% to 80% of patients with AIDS experience anemia, which can be caused by AIDS or by the therapy patients receive for AIDS treatment (for example, AZT). Anemia is a condition in which a patient has below normal levels of hemoglobin, the substance in red blood cells that carries oxygen to all parts of the body. People with severe anemia may experience fatigue and shortness of breath with activity. Therefore, this condition can have a negative influence on a person's quality of life. Epoetin alfa, used to treat anemia, is a genetically engineered form of a natural hormone, erythropoietin, that stimulates red blood cell production. This is a randomized, double-blind (neither the patient nor the physician knows whether the patient is receiving epoetin alfa or placebo), placebo-controlled, parallel group study with an open-label follow-up period that is designed to evaluate the safety and effectiveness of epoetin alfa treatment in patients with AIDS who are being treated with AZT. The study consists of 3 periods: a screening period to determine if patients are eligible for the study, a double-blind period, and an open-label period. Eligible patients will be randomly assigned to one of two groups: a group receiving epoetin alfa 200 U/kg or a group receiving a matching placebo. Patients will be treated with study medication injected under the skin 3 times per week for 12 weeks (or until their hematocrit reaches 38% to 40%). In the open-label period, all patients receive epoetin alfa injected under the skin for up to 6 months. Effectiveness will be determined by the change in hemoglobin and hematocrit (laboratory tests used to evaluate the severity of anemia), transfusion requirements, the patient's quality of life assessment, and the physician's global evaluation of the drug effect. Safety assessments include the incidence and severity of adverse events during the study, and changes in clinical laboratory tests (hematology, biochemistry, and urinalysis), vital signs, electrocardiograms (ECGs), and physical examination findings. The study hypothesis is that AIDS patients who are receiving AZT and who are treated with epoetin alfa will have a lower incident of anemia compared with patients receiving placebo. Double-blind: epoetin alfa (200 U/kg) or placebo given under the skin 3 times a week for 12 weeks or until hematocrit reaches 38% to 40%. Open-label: epoetin alfa 250 U/kg 3 times a week for up to 6 months (once weekly after hematocrit reaches 38% to 40%). Dosage may be adjusted up to 300 U/kg.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a confirmed diagnosis of AIDS, exhibiting signs and symptoms of AIDS characterized by lymphocytopenia (decrease in the number of lymphocytes [cells that are typical elements of lymph tissue] in the blood) as determined by a finding of <1,000 cells/cubic millimeter
* having a documented HIV antibody (either a history of infections due to the patient's impaired resistance or the presence of severe symptoms, such as persistent fever or night sweats associated with significant weight loss)
* receiving AZT therapy of at least 400 mg/day
* having a hematocrit <=30%, and a history of a >=15% decrease in hematocrit since starting AZT therapy, or that the patient has become dependent on transfusions
* clinically stable for at least 1 month before study entry, with a performance score of 0, 1, or 2.

Exclusion Criteria:

* Patients with a history of any important blood disease or clinically significant disease or malfunction of the lungs, heart, hormones, neurological, gastrointestinal, reproductive or urinary systems, which are not caused by the AIDS infection
* having a sudden onset of infections, dementia due to AIDS, uncontrolled high blood pressure, or an iron deficiency
* received androgen therapy within 2 months of study entry
* having anemia caused by other conditions than AIDS or AZT therapy (for example, certain vitamin deficiencies or bleeding from the gastrointestinal tract)
* having a history of seizures, history of cell damage due to chemotherapy within 1 month before study entry, or a history of substance abuse.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Study Completion 1989-08 (Actual)

PRIMARY OUTCOMES:
Change in hemoglobin and hematocrit (laboratory tests used to evaluate the severity of anemia), transfusion requirements, and patient's quality of life assessment.

SECONDARY OUTCOMES:
Adverse events; changes in clinical laboratory tests, vital sign measurements, ECGs, and physical examination findings; and physician's global evaluation of the overall effect of the drug

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: A study to evaluate the safety and effectiveness of epoetin alfa in AIDS (acquired immunodeficiency syndrome) patients with anemia caused both by their disease and by AZT (zidovudine, an antiviral drug) given as treatment for their disease — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=673&filename=CR005842_CSR.pdf